CLINICAL TRIAL: NCT03113747
Title: Safety and Efficacy Evaluation of Tissue Engineered Construct Based on Allogeneic Adipose-derived Multipotent Mesenchymal Stromal Cells and Platelet-poor Plasma Fibrin Hydrogel to Treat the Patients With Burn Wounds
Brief Title: Allogeneic ADSCs and Platelet-Poor Plasma Fibrin Hydrogel to Treat the Patients With Burn Wounds (ADSCs-BWs)
Acronym: ADSCs-BWs
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: A.A. Partners, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-P1
Record Dates: First submitted 2017-03-31; First posted 2017-04-14 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Second- or Third-degree Burns
Keywords: Allogeneic adipose-derived stem cells; burn wounds; wound healing; regeneration; repair; skin tissue engineering
MeSH Terms: conditions — Neoplasm Metastasis; Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ALLO-ASCs (Experimental): The patients receive ALLO-ADSCs. Biological is applied by surface application over perforated (1:3) autologous skin graft following the covering with hypoadhesive bandage. This procedure is carried out twice - once simultaneously with a skin grafting procedure and 2-3 days following autodermoplasty, while bandaging
  Interventions: Biological: ALLO-ASCs
- The standard treatment (No Intervention): All patients will be subjected to standard stepped treatment of burn wounds:
  * Infusion therapy aimed to eliminate disorders of homeostasis during burn shock and burn toxemia;
  * Systemic antibiotic therapy for preventing infectious complications;
  * Adequate analgesia and sedation;
  * Decompression necrotomy in the first 24 hours following the burn trauma;
  * Necrectomy simultaneously with imposition of lyophilized xenografts performed in the first 1-5 days after applying burn;
  * Autologous skin grafting 3-5 days after performed xenografts with the perforation coefficient 1:3

INTERVENTIONS:
Biological: ALLO-ASCs — 1). Cryopreserved cell suspension of early passages of cultured allogeneic MSCs isolated from SVF obtained from lipoaspirate, a total of 10 mln. of cultured cells; 2).The TE-construct consisting of collagen- or fibrin-derived hydrogels and cells of early passages (up to P5) suspension of allogeneic cultured MSCs isolated from SVF obtained from lipoaspirate; Biological is applied by surface application over perforated (1:3) autologous skin graft following the covering with hypoadhesive bandage. This procedure is carried out twice - once simultaneously with a skin grafting procedure and 2-3 days following autodermoplasty, while bandaging.
  Other Names: Allogeneic adipose-derived stem cells
  Arms: ALLO-ASCs

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of tissue engineered construct based on allogeneic cultured adipose-derived multipotent mesenchymal stromal cells (ALLO-ADSCs) and platelet-poor plasma fibrin hydrogel to treat patients with 2-B and 3- degree burn wounds

DETAILED DESCRIPTION:
For more than 20 years in clinical practice allogeneic transplantation of diploid fibroblasts (ADP) for burn wounds has been successfully used, it is used as an independent method, and a method of preparing wounds for autologous skin grafting [1].

The clinical efficacy of transplantation ADP, after the research done by E.V. Glushchenko; Rahayev AM [2,3] is not doubted.

Several studies have shown the efficacy of stem cells in promoting faster and superior wound healing. Alexaki [4] successfully used adipose derived mesenchymal stem cells in wound healing in mice and compared their effect with dermal fibroblasts. The application of stem cells in wounds promoted more efficient reepithelialization by their proliferative effect on keratinocytes.

In recent years, the world's leading burn centers attempted to restore the skin over large areas of burn wounds by epidermal layers transplantation of allogeneic cells cultured in culture medium.

The information expected in the study will be based on the principles of evidence-based medicine and will have practical significance for the treatment of burn wounds.

It is expected to show a positive effect of cultured multipotent mesenchymal stromal cells in the epithelization of burn wounds process as well as the extent and speed healing of skin flap during autologous skin grafting.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18-65 years;
* Patients with 2-nd B and 3-d degree burn wound;
* Body surface area involved in burns - from 10 to 50%;
* The area of skin grafting - less than 6% of the skin surface;
* Burn occurring within the 24 hours prior to the hospitalization;
* Adequate antishock therapy in the prehospital phase;
* Women of childbearing age to provide proof of a current, valid negative pregnancy test;
* Confirmation of participation in the study by signing the Instrument of Consent, personally or through a responsible caretaker.

Exclusion Criteria:

* Prognostically favorable or unfavorable outcome of the disease
* (Lesion Severity Index, less than 30 or more, than 120 score);
* Combined trauma;
* Severe respiratory tract burn injuries;
* Ischemic disease of the lower extremities;
* The presence of cardiovascular disease (CVD): symptoms of unstable angina, myocarditis, heart disease, heart failure;
* History of prior cancer;
* Healing of duodenal or gastric ulcers in history;
* Diabetes
* Severe chronic liver diseases or kidney disease in history;
* History of alcohol or other drug abuse;
* Pregnanсy;
* Any other physical diseases in decompensation or subcompensation,
* or those that are rated as severe or moderate;
* Therapeutic issues or psychiatric disorders of a patient which would
* make the subject unsuitable to participate in this study or to complete it;
* Participation in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03-25 (Actual); Primary Completion 2018-12-26 (Estimated); Study Completion 2018-12-26 (Estimated)

PRIMARY OUTCOMES:
The degree of healing of skin flap; The degree of epithelialization of burn wounds in the perforations of a skin graft | up to 1 month
  The degree of healing of skin flap after autologous skin grafting;

SECONDARY OUTCOMES:
The dynamics of healing of skin flap | up to 1 month
  Complete epithelization or epithelization more than 50% of the cells in the skin graft on the 10th day after autologous skin grafting are effective. The epithelialization less than 50% is not effective.
Dynamics of the phagocytic activity of neutrophils in the area of burn wounds, according to NBT-test. | up to 1 month
  Dynamics of the phagocytic activity of neutrophils in the area of burn wounds, according to NBT-test.
Duration of treatment (days) to complete epithelialization of burn wounds; | up to 1 month
  Duration of treatment (days) to complete epithelialization of burn wounds;

CONTACTS AND LOCATIONS:
Overall Officials: Anatoliy V. Voronin, Principal Investigator — The head doctor of The Kyiv City Clinical Hospital №2; Georgiy P. Kozynets, MD, PhD, DSc, Principal Investigator — Head of the department of combustiology and plastic surgery, Shupyk National Medical Academy of Postgraduate Education
Locations (1):
- The Kyiv City Clinical Hospital №2, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alexaki VI, Simantiraki D, Panayiotopoulou M, Rasouli O, Venihaki M, Castana O, Alexakis D, Kampa M, Stathopoulos EN, Castanas E. Adipose tissue-derived mesenchymal cells support skin reepithelialization through secretion of KGF-1 and PDGF-BB: comparison with dermal fibroblasts. Cell Transplant. 2012;21(11):2441-54. doi: 10.3727/096368912X637064. Epub 2012 Apr 10. PMID 22507764
- See also: Adipose tissue-derived mesenchymal cells support skin reepithelialization through secretion of KGF-1 and PDGF-BB: comparison with dermal fibroblasts. — https://www.ncbi.nlm.nih.gov/pubmed/22507764
- See also: 2. Allografting of cultured fibroblasts on nonhealing wounds after autodermoplasty. D. S. Sarkisov, E. V. Glushchenko, Sh. R. Gurukov, S. S. Morozov, V. P. Tumanov, N. V. Berezhkov Bulletin of Experimental Biology and Medicine/May 1991, Volume 111, Issue — http://www.fesmu.ru/elib/Article.aspx?id=60810
- See also: 3. Alekseev AA, Krutikov MG, Rakhaev AM/ Treatment of border burns and donor wounds with cultured allofibroblasts// Annals of Surgery. 2001. № 1. С. 59-65. — http://www.fesmu.ru/elib/Article.aspx?id=60810
- See also: 4. Alexaki V.-I. et al. Adipose tissue-derived mesenchymal cells support skin reepithelialization through secretion of KGF-1 and PDGF-BB: comparison with dermal fibroblasts. Cell Transplantation. 2012;21(11):2441-2454. — https://www.ncbi.nlm.nih.gov/pubmed/22507764